CLINICAL TRIAL: NCT00226005
Title: Phase II Trial of PTK787/ZK222584 in Patients With Advanced or Metastatic Pancreatic Adenocarcinoma Who Failed First-Line Gemcitabine Therapy.
Brief Title: PTK787 in Patients With Advanced Metastatic Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pancreatic Cancer Research Team (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCRT04-001
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Neoplasm
Keywords: pancreas; adenocarcinoma; cancer; metastatic; advanced cancer; Phase II; growth factor; VEGF; angiogenesis
MeSH Terms: conditions — Neoplasms; Adenocarcinoma; Neoplasm Metastasis | interventions — vatalanib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vatalanib (Active Comparator): Administered orally, twice daily: after enrollment - first week 250 BID, second week 500 BID, then 750 BID thereafter.
  Interventions: Drug: PTK787/ZK222584

INTERVENTIONS:
Drug: PTK787/ZK222584 — One arm: administered orally, twice daily: after enrollment - first week 250 BID, second week 500 BID, then 750 BID thereafter.
  Other Names: bevacizumab

SUMMARY:
The purpose of this research study is to find out if an experimental drug called PTK787/ZK222584 might be effective against advanced or metastatic pancreatic cancer.

In order for tumors to grow and spread to other parts of the body, they need to have a growing blood supply. Tumor cells have been shown to produce substances that stimulate the abnormal growth of new blood vessels that allow the tumor to grow. In adults, blood vessel cells normally divide very rapidly. It is thought that PTK787/ZK222584 may interfere with the growth of new blood vessels. A drug that interferes with the growth of new blood vessels might stop tumor growth, and possibly shrink the tumor by keeping it from receiving nutrients and oxygen supplied by the blood vessels. Since normal blood vessel cells divide very rarely, it might be possible to stop tumor growth without harming normal tissues.

DETAILED DESCRIPTION:
This is an open-label, phase II multi-center therapeutic trial investigating the efficacy and tolerability of PTK787/ZK222584 in patients with metastatic or advanced pancreatic cancer who failed first line gemcitabine-based therapy. The primary objective of this study is to evaluate the 6-month survival rate, time to progression, and tolerability of the regimen in pancreatic cancer patients treated with PTK787/ZK222584 as second-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Zubrod performance status of 0 - 2
* Histological or cytological diagnosis of pancreatic adenocarcinoma
* Measurable or evaluable disease determined as per RECIST criteria
* Life expectancy > 12 weeks
* Written informed consent
* Patients must have failed or progressed on prior gemcitabine-based therapy for advanced or metastatic disease.

Exclusion Criteria:

* Islet cell or neuroendocrine carcinomas of the pancreas.
* History or presence of central nervous system disease.
* Patients with a history of another primary malignancy < 5 years
* Prior chemo therapy < 21 days prior to registration.
* Prior biologic or immunotherapy < 14 days prior to registration
* Prior full field radiotherapy < 28 days or limited field radiotherapy < 14 days prior to registration.
* Major surgery < 28 days prior to registration.
* Patients who have received investigational drugs < 28 days prior to registration.
* Prior therapy with anti-VEGF agents.
* Pleural effusion or ascites that causes respiratory compromise.
* Female patients who are pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2005-12; Primary Completion 2008-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the 6-month survival rate and time to progression in pancreatic cancer patients treated with PTK787/ZK222584. | DSMC Schedule
  The Data Safety Monitoring Board met twice yearly while the study was active (2006-2008) to review data and each of the primary and secondary objectives.
  Safety Issue: the only endpoint/outcome measure that was a safety issue was the second one (safety and tolerability of PTK)

SECONDARY OUTCOMES:
To assess the response rates of patients treated with PTK787/ZK222584. | DSMC Schedule
  The Data Safety Monitoring Board met twice yearly while the study was active (2006-2008) to review data and each of the primary and secondary objectives.
To evaluate DCE-MRI as a surrogate of response to PTK787/ZK222584 therapy in pancreatic cancer patients. | DSMC Schedule
  The Data Safety Monitoring Board met twice yearly while the study was active (2006-2008) to review data and each of the primary and secondary objectives.
To perform analysis of tissue, blood and plasma markers that may be helpful in assessing the likelihood of benefit from PTK787/ZK222584 therapy. | DSMC Schedule
  The Data Safety Monitoring Board met twice yearly while the study was active (2006-2008) to review data and each of the primary and secondary objectives.

CONTACTS AND LOCATIONS:
Overall Officials: Tomislav Dragovich, MD, PhD, Principal Investigator — University of Arizona/Arizona Cancer Center
Locations (7):
- United States (7):
  - Scottsdale Healthcare, Scottsdale, Arizona
  - University of Arizona/Arizona Cancer Center, Tucson, Arizona
  - Tower Hematology Oncology Medical Group, Beverly Hills, California
  - Sidney Kimmel Comprehensive Cancer Center/Johns Hopkins, Baltimore, Maryland
  - Virginia Piper Cancer Institute/Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - South Texas Oncology and Hematology, San Antonio, Texas

REFERENCES:
- See also: web page for the nonprofit group, Pancreatic Cancer Research Team — http://www.pcrt.org